CLINICAL TRIAL: NCT05733117
Title: Supplementation Efficacy Comparing the Oral Nano and Conventional Vitamin D in Inflammatory Bowel Disease
Brief Title: Oral Nano Vitamin D Supplementation Efficacy in Inflammatory Bowel Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tomas Bata Hospital, Czech Republic (Other)
Collaborators: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Vladimir Kojecky, MD, Ph.D., Head of dept. of internal medicine, Tomas Bata Hospital, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K092022
Record Dates: First submitted 2022-09-25; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Vitamin D Substitution
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NanoVitD (Active Comparator): Oral nano form of the calciferol
  Interventions: Drug: Vitamin D
- ConvVitD (Active Comparator): Conventional oral calciferol
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — cholecalciferol

SUMMARY:
The purpose of this study is to compare efficacy of the suplementation using the conventional oral and oral nano form of the calciferol.

DETAILED DESCRIPTION:
Conventional oral vit D formulas have variable availability esp. in IBD patients. Oral nano vitamin D is absorbed in the mouth. The aim of this study is to compare the efficacy of both formulations by matching vitD levels after supplementation and to determine the equivalent dose.

ELIGIBILITY:
Inclusion Criteria:

* The inflammatory bowel disease patients

Exclusion Criteria:

* Liver and renal disease
* Hypercalcemia
* Hyperparathyreoidism
* Chronic pancreatitis
* Concomitant vitamin D medication
* Pregnancy
* Sarcoidosis
* Malignancy
* Inability to obtain valid data from subject

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Vitamin D (25OHD) blood level | 4 months
  Change of the D vitamin level after follow-up interval

CONTACTS AND LOCATIONS:
Overall Officials: Vladimír Kojecký, MD, Principal Investigator — Tomas Bata Hospital, Czech Republic
Locations (2):
- Czechia (2):
  - Faculty Hospital Kralovske Vinohrady, Prague
  - ThomasBH, Zlín

IPD SHARING:
Plan to Share IPD: No